CLINICAL TRIAL: NCT03262129
Title: Type 1 Multiple Endocrine Neoplasia : a Cohort Study of the Endocrine Tumor Study Group (GTE)
Brief Title: Type 1 Multiple Endocrine Neoplasia Cohort Study
Acronym: MEN1-GTEcohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GOUDET PARI 2011
Record Dates: First submitted 2016-08-31; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Type 1-Multiple Endocrine Neoplasia Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Type 1 - Multiple Endocrine Neoplasia syndrome (MEN1,) is an autosomal dominant disorder secondary to MEN1 mutations that predisposes carriers to endocrine tumors. The MEN1 gene located on chromosome 11q13 encodes menin, a 610 amino acid protein expressed in all tissues tested. Menin is a scaffold protein which interacts with a large number of intracellular molecules. MEN1 disease may display various clinical associations The tumors mainly develop from endocrine tissues and may arise from parathyroid glands, duodeno-pancreas, pituitary gland, adrenal glands, and at a lower frequency from the bronchi and thymus. The penetrance is very progressive but ultimately high during a lifespan.

Although the syndrome was discovered in 1903 by Erdheim and properly documented in 1954 by Wermer, it was only in the 1970s that the variety of clinical presentations was acknowledged and first attempts to codify treatments were made. Most published studies deals with selected and small size populations. Thus, many aspects of the natural history of MEN1 remains unknown as well as the optimal care of patients. In addition, although advances in genetics improved the diagnosis of MEN1, there are still clinical forms whose attachment to the syndrome is difficult: atypical, paucisymptomatic, forms the negative genetic diagnosis (10%). These clinical forms need to be clarified to ensure optimum support.

This cohort relies on the Groupe d'étude des Tumeurs Endocrines (GTE) network for MEN1, created in February 1991, and brings together clinical centers in France and Belgium (n=80) as well as the four genetics laboratories in charge of MEN1 diagnosis. It aims at improving the knowledge of the MEN1mainly in describing:

* its evolution over time globally and according to the initial presentation, ( particularly accounting the risk of the occurrence of secondary MEN1 related or unrelated tumors, and death)
* the genotype-phenotype correlations and heritability of the disease
* the real life management of patients and its impact on cure and survival for each type of MEN1-related tumor
* the impact of the NEM on the patients' daily lives, their perception of the disease and their satisfaction with their care

ELIGIBILITY:
Patients with MEN1 according to the Gubbio criteria :

* Patients with a MEN1 mutation and presenting at least one of the following symptomatic or silent lesions: pHPT or pancreatic or duodenal endocrine tumor
* Pituitary tumor
* Adrenal tumor
* th-NET
* br-NET
* And gastric enterochromaffin-like tumor (ECLoma).
* Patients belonging to a known MEN1 family (at least one first-degree relative affected) and presenting at least one of the aforementioned lesions.
* Patients without positive genetic testing or a family background presenting at least two of the three major MEN1 lesions (pHPT, pancreatic, or duodenal endocrine tumor, pituitary tumor).:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Vital status | 12 months
MEN-1 related tumors | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France